CLINICAL TRIAL: NCT01536080
Title: Comparison of Risk Factors, GERD Symptoms and PPI Responses in the Reflux Esophagitis, Non-erosive Reflux Disease and Functional Heartburn Using GERD Impact Scale Questionnaire
Brief Title: Analysis of GERD Symptoms Using Gastroesophageal Reflux Impact Score Questionnaire for Quality of Life
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, M.D., Seoul National University Bundang Hospital
Other Study IDs: D9612L00150
Record Dates: First submitted 2012-02-13; First posted 2012-02-20 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Reflux Esophagitis (RE); Non-erosive Reflux Disease (NERD); Functional Heartburn (FH)
MeSH Terms: conditions — Esophagitis, Peptic; Non-Erosive Reflux Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Reflux esophagitis (RE)
- Non-erosive reflux disease (NERD)
- Functional heartburn (FH)

SUMMARY:
Even the patients complain GERD symptoms such as heartburn and acid regurgitation the final diagnosis could be reflux esophagitis (RE), non-erosive reflux disease (NERD) and even functional heartburn (FH). In addition, the GERD symptoms are consisted of esophageal symptoms and extraesophageal symptoms. Thus it is necessary to use effective tool for the measurement of GERD symptoms and response of proton pump inhibitor in short time. Several questionnaires have been made for the assessment of GERD symptoms in recent years However, their screening tools do not include the impact of symptoms on everyday life and take a long time to complete the questionnaires. The GERD impact scale (GIS) questionnaire has been developed to compensate for this. It is a simple, one-page, questionnaire to communicate to the doctor the frequency of reflux symptoms and their effect on quality of life, recognizing that it might also prompt clinicians to make appropriate treatment for patients' symptoms. However, there was no report regarding comparison of the characteristics and response to PPI in RE, NERD and FH groups using GIS questionnaire so far.

ELIGIBILITY:
Inclusion Criteria:

* Adult Subjects (From 16 to 85 years old)
* The subjects with GERD symptom who received 8 week PPI therapy

Exclusion Criteria:

* Patients with a history of gastrointestinal surgery, Barrett's esophagus, esophageal motility disorder, duodenal ulcer, benign gastric ulcer or gastroduodenal cancer and systemic disease requiring chronic medication (except for hypertension and diabetes mellitus)
* Patients who took H2 blocker or a PPI to relieve these symptoms within 4 weeks

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Even the patients complain GERD symptoms such as heartburn and acid regurgitation the final diagnosis could be reflux esophagitis (RE), non-erosive reflux disease (NERD) and even functional heartburn (FH).
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2008-07

PRIMARY OUTCOMES:
The GIS score at baseline | Before 8 weeks PPI treatment(baseline)

SECONDARY OUTCOMES:
Change of the GIS score from baseline | After 8 weeks PPI treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Bundang-gu, Seongnam, Gyeonggi-do, South Korea